CLINICAL TRIAL: NCT05779137
Title: The Effect of Mindfulness-based Cognitive Therapy on Psychological Distress in People With Parkinson's Disease
Brief Title: The Effects of Mindfulness-based Cognitive Therapy in People With Parkinson's Disease
Acronym: MIND-PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: NL81309.091.22
Record Dates: First submitted 2023-01-12; First posted 2023-03-22 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Mindfulness; Mindfulness-based cognitive therapy; Disease progression
MeSH Terms: conditions — Parkinson Disease; Disease Progression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The involved researchers will not be blinded to the treatment allocation, because this would not be feasible with the current design. Patients receiving MBCT need to be allocated to a specific treatment group, which requires extensive communication between the patient, mindfulness center and researcher. Also, patients receiving the treatment will perform different questionnaires in the course of the study, which makes it impossible for the researcher to be blinded for group allocation. We do not expect any bias on our primary outcome measure (self-report questionnaire). Secondary outcome measures (MRI, blood serum, hair cortisol) are unlikely to be biased by the researcher. UPDRS-III performance will be video recorded to allow blinded ratings by independent researchers after collecting the data (hence blinded outcome assessor). Patients will be informed about their intervention after randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness based cognitive therapy (MBCT) (Experimental): 62 patients will receive a mindfulness based intervention.
  Interventions: Behavioral: MBCT
- Treatment as usual (TAU) (No Intervention): 62 patients will receive treatment as usual, this will form a (passive) control group to the MBCT group.
- Healthy control (HC) (No Intervention): 50 healthy individuals without PD will not be randomized. This arm will only be measured once at baseline.

INTERVENTIONS:
Behavioral: MBCT — Patients will join a mindfulness-based cognitive therapy course at the Radboudumc Center for Mindfulness. The course consists of eight weekly sessions of 2.5-hour and one 6-hour silence day between the 6th and 7th session. The sessions include meditation exercises (body-scan, sitting meditation, gentle movement exercises, three-minute breathing space, daily activities with attention), psychoeducation and group discussion. Psychoeducation includes information on cognitive techniques, like monitoring and scheduling of events and identification of negative automatic thoughts. In addition, all participants will be encouraged to perform daily practice assignments at home for about 30-45 minutes per day, mainly consisting of meditation exercises.
  Arms: Mindfulness based cognitive therapy (MBCT)

SUMMARY:
Parkinson's disease (PD) is a debilitating neurodegenerative disorder occurring in 7 million patients worldwide. PD is caused by progressive loss of nigro-striatal dopamine cells, which causes motor symptoms such as slowness of movement and tremor, and non-motor symptoms such as cognitive dysfunction. Converging clinical evidence indicates that PD patients are very sensitive to the effects of psychological stress. There is a high prevalence of stressrelated neuropsychiatric symptoms in PD: 30-40% of patients experience depression and 25-30% have anxiety. Furthermore, stress worsens many motor symptoms, e.g. tremor, freezing of gait, and dyskinesia. In addition to these immediate negative effects, chronic stress may also have detrimental long-term consequences, and specifically by accelerating disease progression, as suggested by animal models. However, this hypothesis remains to be confirmed in humans. Better evidence about the impact of stress on PD would have major treatment consequences: novel stress-reducing interventions may have symptomatic effects, and perhaps also disease-modifying effects. The aim of this study is to test whether a stress-reducing intervention improves clinical symptoms, slows neurodegeneration, and/or enhances neuroplasticity in PD. In a randomized controlled trial, the investigators will compare a stress-reducing mindfulness-based intervention group (MBI; one year) to a treatment as usual (TAU) group on clinical symptoms, cerebral markers of nigro-striatal dysfunction and stressor-reactivity (MRI), and inflammatory markers (serum).

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a common and fast-growing neurological disease, clinically characterized by motor slowing (bradykinesia), stiffness (rigidity) and resting tremor. The pathological hallmark of PD is nigro-striatal dopamine depletion, but the noradrenergic (stress) system is also affected. Indeed, the prevalence of stress-related neuropsychiatric symptoms in PD is high and many PD patients suffer from reduced health-related quality of life. Also, (chronic) stress worsens many motor symptoms and may have detrimental long-term consequences by accelerating disease progression, as suggested by animal models.

There is no cure for PD, and currently no treatments to slow down disease progression. Therefore, the development of new and effective treatments is crucial. Given the large role of stress on PD symptoms, stress reduction might improve motor as well as non-motor symptoms. Intriguingly, recent evidence suggests that mindfulness training, where mindfulness is the trainable capacity to experience the present moment on purpose and without judgment, is an effective way to achieve such stress reduction. In fact, the effects of mindfulness practice have gained much interest as a topic of scientific research and clinical practise recently, where Mindfulness-Based Cognitive Therapy (MBCT) is one of the most commonly applied interventions, shown to be effective for a variety of somatic and psychiatric disorders. Importantly, previous trials investigating the effect of mindfulness-based interventions (MBIs) on clinical symptoms in PD showed positive effects on depression in 6/8 trials, on anxiety in 4/7 trials and on motor symptoms in 2/3 studies. Also, a large online survey on patients' experiences with stress and mindfulness showed that on one hand, patients experienced considerably more stress than controls, and significant stress-related worsening of PD symptoms; on the other, PD mindfulness users reported positive effects of mindfulness on anxiety and depression. In summary, current evidence suggests a positive effect of MBIs on psychological distress in PD, but clinical evidence is inconclusive. Also, to date, there is no research on the (cerebral) mechanisms underlying the (positive) effects of mindfulness in PD. Insight to the cerebral mechanisms of MBIs can pave the way for developing new, mechanism-based interventions, and can help to uncover the nature of the effects of stress on Parkinson's disease. Specifically, a mechanism based approach allows us to disentangle the symptomatic (stress as an amplifying factor on motor dysfunction) as opposed to neurodegenerative (nigro-striatal cell loss) effects of stress.

In this study, the investigators will test the effect of MBCT on the clinical (symptomatic) and neurodegenerative course of PD. If proven to be effective, MBCT can be applied as a new and cost-effective therapy to PD patients. The investigators will perform a randomized controlled trial with MBCT as intervention and a treatment as usual (TAU) control group. The investigators will evaluate whether a MBCT mindfulness course can lead to clinically relevant reductions in psychological distress (measured with the Hamilton Anxiety and Depression Scale) in PD patients with mild to moderate symptoms of psychological distress. Also, the investigators will evaluate the effects of a MBCT mindfulness course on other PD symptoms (e.g. motor dysfunction), cerebral markers of neurodegeneration, and neuroplasticity, and explore whether the intervention lowers systemic inflammatory tone in PD. The total duration of data acquisition per participant will be 12 months, consisting of a baseline measurement (T0), an intervention period of 2 months followed by a post-measurement (T1), and a final measurement (T2) that takes place 12 months after T0.

ELIGIBILITY:
Inclusion criteria for the RCT:

* A diagnosis of idiopathic PD made by a movement disorders specialist.
* PD disease duration is ≤10 years, defined as time since diagnosis made by a neurologist.
* Mild-moderate symptoms of psychological distress (Hospital Anxiety and Depression Scale score >10 points).
* Subject can read and understand the Dutch language.

Exclusion criteria for the RCT:

* Severe neurological or psychiatric co-morbidity (e.g. psychosis or suicidality).
* Contraindications for MRI (e.g. brain surgery in medical history, claustrophobia, an active implant, epilepsy, pregnancy, and/or metal objects in the upper body that are incompatible with MRI).
* Moderate to severe head tremor (to avoid artifacts caused by extensive head motion during scanning).
* Cognitive dysfunction (clinical diagnosis of dementia, or a score of 20 or lower on the MoCA, which will be measured at T0).
* Previous participation in MBSR or MBCT (>4 sessions).

Inclusion criteria (HC group):

• Participants of the HC group must be able to read and understand the Dutch language.

Exclusion criteria (HC group):

* Severe neurological or psychiatric co-morbidity (e.g. psychosis or suicidality).
* Contraindications for MRI (e.g. brain surgery in medical history, claustrophobia, an active implant, epilepsy, pregnancy, and/or metal objects in the upper body that are incompatible with MRI).
* Cognitive dysfunction (clinical diagnosis of dementia, or a score of 20 or lower on the MoCA, which will be measured at T0).
* Detailed knowledge about the nature of the stress induction paradigm prior to participating in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Psychological distress post-intervention (as assessed by HADS [0-42]) | Month 2
  Our primary outcome will be psychological distress (anxiety and depressive symptoms), measured by the Hospital Anxiety and Depression Scale (HADS) at T1 (post-intervention). The HADS is a validated self-report questionnaire consisting of anxiety and depression subscales, scores can range from 0-42 points. Lower scores mean less stress, i.e. better outcome. It was previously used as primary outcome measure in an MBCT-RCT in cancer, it was used as outcome measure in the largest MBI-RCT to date in PD, and it has been validated in PD.
  The effect on HADS will all be analyzed with an analysis of covariance (ANCOVA). The dependent variable will be the HADS score at T1; group allocation will serve as fixed factors, and age at T0, sex and the HADS score at T0 will serve as covariates.

SECONDARY OUTCOMES:
Change in psychological distress (as assessed by HADS [0-42]) | Month 12. Change relative to baseline.
  HADS [0-42] (lower score = better (less stress), see also primary outcome.
Disease severity (as assessed by MDS-UPDRS [0-199]) | Month 0, month 2, month 12.
  MDS-UPDRS [0-199] (higher score = worse (more disability)). We will assess overall symptom severity as a function of time T0/T1/T2 and group (MBCT vs. TAU).
Cognitive function (as assessed by MoCA [0-30]) | Month 0, month 2, month 12.
  Montreal Cognitive Assessment; MoCA [0-30] (higher score = better (less disability)) We will test whether clinical scores change significantly between T0, T1 and T2 using mixed models.
Tremor severity (indicated by tremor power [log(µV2)]) | Month 0, month 2, month 12.
  We will compare tremor severity as measured with accelerometry during rest, mental arithmetic (coco), posturing and action. We will perform a 2x2x2 ANOVA with between-subjects factor GROUP (MBCT vs. control), and within-subjects factors TIME (T0 vs. T2) and CONDITION (coco vs. rest, posture vs. rest, action vs. rest).
Hair cortisol | Month 0, month 2, month 12.
  Hair cortisol levels will be established by means of a hair sample and hair cortisol concentration of the previous 2 months will be assessed and compared between T0/T1/T2 and between groups (MBCT/TAU)
Bradykinesia severity (indicated by average keys per second on key tapping test) | Month 0, month 2, month 12.
  We will measure bradykinesia severity by means of a keyboard finger tapping test. Average keys pressed per seconds will be used as dependent variable. More keys per second = less disability. We will test whether clinical scores change significantly between T0, T1 and T2 using mixed models.
Inflammatory tone (as assessed by serum C-reactive protein) | Month 0, month 2, month 12.
  We will be assessing inflammatory tone by means of serum C-reactie protein (CRP) levels. Higher CRP = more inflammation.
Quality of life questionnaire (as assessed by PDQ-39 [0-100]) | Month 0, month 2, month 6, month 12.
  Parkinson Disease Questionnaire 39; PDQ-39 [0 - 100] (higher score = worse (more disability)) We will test whether clinical scores change significantly between T0, T1 and T2 using mixed models.
Perceived stress (as assessed by PSS [0-40]) | Month 0, month 2, month 6, month 12.
  Perceived Stress Scale; PSS [0 - 40] (higher score = worse (more perceived stress)) We will test whether clinical scores change significantly between T0, T1 and T2 using mixed models.
Rumination (as assessed by RRS [26-104]) | Month 0, month 2, month 6, month 12.
  Ruminative Response Scale; RRS [26-104] (higher score = worse (more ruminative thoughts)) We will test whether clinical scores change significantly between T0, T1 and T2 using mixed models.
Mindfulness skills (as assessed by FFMQ [39-195]) | Month 0, month 2, month 6, month 12.
  Five Facet Mindfulness Questionnaire Short Form; FFMQ [39-195] (higher score = better (more mindfulness skills)) We will test whether clinical scores change significantly between T0, T1 and T2 using mixed models.
Self-compassion as assessed by SCS [12-84]) | Month 0, month 2, month 6, month 12.
  Self-Compassion Short Form; SCS [12-84] (higher score = better (more self compassion)) We will test whether clinical scores change significantly between T0, T1 and T2 using mixed models.
Self-efficacy (as assessed by GSES [10-40]) | Month 0, month 2, month 6, month 12.
  General Self-Efficacy Scale; GSES [10-40] (higher score = better (more self efficacy)) We will test whether clinical scores change significantly between T0, T1 and T2 using mixed models.
Positive appraisal (as assessed by PASS) | Month 0, month 2, month 6, month 12.
  Positive Appraisal Style Scale; PASS [for each coping style: 2-10, for humor: 1-8] We will test whether clinical scores change significantly between T0, T1 and T2 using mixed models.
Decision making task | Month 0, month 2, month 12.
  Patients will perform a neuropsychological task designed to track individual decision making and learning processes. Computational modeling will be used to model response patters according to an actor model and a spectator model. Response patterns will be compared as a function of group (MBCT / TAU) and time (T0 / T1/ T2).
Salivary cortisol | Month 0, month 12.
  Acute cortisol levels will be assessed via saliva samples during socially evaluated cold pressor test as a function of group (MBCT/TAU), time (T0/T2), and SECPT time points (pre/post/30mpost/60mpost).
Resting state network reactivity to a stressor (fMRI) | Month 0, month 12.
  Resting-state network connectivity will be assessed based on resting state fMRI before and after the socially evaluated cold pressure test (SECPT). In specific, this will be evaluated as a function of group (MBCT / TAU), time (T0 / T2), and SECPT (before / after). Resting state networks of interest include the salience network, central executive network, and default mode network.
Grey matter volume of stress-related regions (MRI) | Month 0, month 12.
  By means of a structural T1 scan, we will compare structural changes in stress-related brain regions, e.g. amygdala, hippocampus. Specifically, grey matter volume will be compared as a function of group (MBCT / TAU) and time (T0 / T2).
  This measure will help us distinguish between structural changes versus network adaptations as a response to the intervention.
Structural integrity of substantia nigra and locus coeruleus (LC) | Month 0, month 12.
  To further evaluate structural integrity of the substantia nigra and LC, signal intensity on neuromelanin sensitive MRI scans, as well as diffusion MRI will be determined before and one year after the MBI. Structural integrity will be analysed as a function of group (MBCT / TAU) and time (T0 / T2).
Functional integrity of nigro-striatal dopamine system | Month 0, month 12.
  To quantify the functional integrity of the nigro-striatal dopamine system, we will use resting-state fMRI to calculate gradients of cortico-striatal connectivity. This fMRI measure is sensitive to compensatory changes: in PD, cortico-striatal connectivity shifts from more-affected (posterior) to less-affected (anterior) portions of the striatum. To investigate this, functional connectivity profiles of the posterior and anterior putamen specifically will be determined and analysed as a function of group (MBCT / TAU) and time (T0 / T2).
Hair cortisol (HC) | Month 0
  Hair cortisol levels will be established by means of a scalp hair sample. Hair cortisol concentration of the previous 3 months will be assessed and compared between groups (PD/HC).
Decision making task (HC) | Month 0
  Patients will perform a neuropsychological task designed to track individual decision making and learning processes. Computational modeling will be used to model response patterns according to an actor model and a spectator model. Response patterns will be compared as a function of group (PD/HC).
Salivary cortisol (HC) | Month 0
  Acute cortisol levels will be assessed via saliva samples during socially evaluated cold pressor test as a function of group (PD/HC) and SECPT time points (pre/post/30mpost/60mpost).
Resting state network reactivity to a stressor (fMRI) (HC) | Month 0
  Resting-state network connectivity will be assessed based on resting state fMRI before and after the socially evaluated cold pressor test (SECPT). In specific, this will be evaluated as a function of group (PD/ HC) and SECPT (before / after). Resting state networks of interest include the salience network, central executive network, and default mode network. Relevant mediators of the effect will be explored.
Structural integrity of substantia nigra and locus coeruleus (HC) | Month 0
  To evaluate structural integrity of the substantia nigra and locus coeruleus, signal intensity on neuromelanin sensitive MRI scans, as well as diffusion MRI will be determined. Structural integrity will be analysed as a function of group (PD/ HC).

CONTACTS AND LOCATIONS:
Overall Officials: Rick Helmich, MD PhD, Principal Investigator — Radboud University Medical Centre; Donders Institute for Brain, Cognition and Behaviour
Locations (1):
- Donders Centre for Cognitive Neuroimaging, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cieza A, Causey K, Kamenov K, Hanson SW, Chatterji S, Vos T. Global estimates of the need for rehabilitation based on the Global Burden of Disease study 2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2021 Dec 19;396(10267):2006-2017. doi: 10.1016/S0140-6736(20)32340-0. Epub 2020 Dec 1. PMID 33275908
- [Background] Kish SJ, Shannak K, Hornykiewicz O. Uneven pattern of dopamine loss in the striatum of patients with idiopathic Parkinson's disease. Pathophysiologic and clinical implications. N Engl J Med. 1988 Apr 7;318(14):876-80. doi: 10.1056/NEJM198804073181402. PMID 3352672
- [Background] Hemmerle AM, Herman JP, Seroogy KB. Stress, depression and Parkinson's disease. Exp Neurol. 2012 Jan;233(1):79-86. doi: 10.1016/j.expneurol.2011.09.035. Epub 2011 Oct 6. PMID 22001159
- [Background] van der Heide A, Speckens AEM, Meinders MJ, Rosenthal LS, Bloem BR, Helmich RC. Stress and mindfulness in Parkinson's disease - a survey in 5000 patients. NPJ Parkinsons Dis. 2021 Jan 18;7(1):7. doi: 10.1038/s41531-020-00152-9. PMID 33462213
- [Background] de Pablos RM, Herrera AJ, Espinosa-Oliva AM, Sarmiento M, Munoz MF, Machado A, Venero JL. Chronic stress enhances microglia activation and exacerbates death of nigral dopaminergic neurons under conditions of inflammation. J Neuroinflammation. 2014 Feb 24;11:34. doi: 10.1186/1742-2094-11-34. PMID 24565378
- [Background] Burtscher J, Copin JC, Rodrigues J, Kumar ST, Chiki A, Guillot de Suduiraut I, Sandi C, Lashuel HA. Chronic corticosterone aggravates behavioral and neuronal symptomatology in a mouse model of alpha-synuclein pathology. Neurobiol Aging. 2019 Nov;83:11-20. doi: 10.1016/j.neurobiolaging.2019.08.007. Epub 2019 Aug 14. PMID 31585362
- [Background] van der Heide A, Meinders MJ, Speckens AEM, Peerbolte TF, Bloem BR, Helmich RC. Stress and Mindfulness in Parkinson's Disease: Clinical Effects and Potential Underlying Mechanisms. Mov Disord. 2021 Jan;36(1):64-70. doi: 10.1002/mds.28345. Epub 2020 Oct 23. PMID 33094858
- [Background] Baer, R. A. Mindfulness training as a clinical intervention: a conceptual and empirical review. Clinical psychology: Science and practice 10, 125-143, doi:10.1093/clipsy.bpg015 (2003).
- [Derived] van der Heide A, Goltz F, de Vries NM, Bloem BR, Speckens AE, Helmich RC. Study protocol for the MIND-PD study: a randomized controlled trial to investigate clinical and biological effects of mindfulness-based cognitive therapy in people with Parkinson's disease. BMC Neurol. 2024 Jun 25;24(1):219. doi: 10.1186/s12883-024-03736-7. PMID 38918695

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-25): https://cdn.clinicaltrials.gov/large-docs/37/NCT05779137/Prot_SAP_000.pdf